CLINICAL TRIAL: NCT03300765
Title: Intensity Modulated Radiation Therapy Combined With Apatinib for Inoperable or Iodine Refractory Thyroid Cancer: A Phase II Single-arm Study
Brief Title: Trail Evaluating Apatinib With IMRT for Inoperable or Iodine Refractory Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiayun He, MD (Other)
Responsible Party: Sponsor-Investigator, Xiayun He, MD, Chief Physician, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-Shanghai
Record Dates: First submitted 2017-09-26; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; Apatinib; Intensity modulated radiation therapy
MeSH Terms: conditions — Thyroid Neoplasms | interventions — apatinib; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib with IMRT (Experimental): Participants will receive apatinib (0.5g, daily) for two cycles followed by intensity modulated radiation therapy (Primary site and lymph nodes: 66 Gy/33F, metastatic site: 40-60Gy/20-30F)
  Interventions: Drug: Apatinib; Radiation: Intensity modulated radiation therapy

INTERVENTIONS:
Drug: Apatinib — Apatinib will be used as induction therapy in experimental arm.
Radiation: Intensity modulated radiation therapy — Intensity modulated radiation therapy will be used for patients with progression disease during induction therapy or after induction therapy.

SUMMARY:
To determine the efficacy and safety of intensity modulated radiation therapy combined with apatinib for inoperable or iodine refractory thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand character and individual consequences of the clinical trial. Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial;
* Aged ≥ 18 years old;
* Pathologically confirmed inoperable or iodine refractory thyroid cancer, or postoperative residual disease detected by imaging studies, or progression disease within 12 months before enrollment. (all with measurable disease ≥10mm according to RECIST 1.1);
* ECOG0-2;
* Adequate laboratory values within 14 dyas of enrollment to study defined as follows: N ≥ 1500/mm^3; PLT ≥ 80,000/mm^3; HB≥90g/L;total bilirubin < 1.25ULN; AST/ALT < 2.5 ULN or < 5 ULN with metastasis; SCr ≤1ULN; CCR > 50ml/min;
* The survival period is expected to be greater than 3 months;
* Willing to accept adequate contraception for patients with childbearing potential.

Exclusion Criteria:

* Take chemotherapeutic chemotherapy (the use of low-dose chemotherapy for radiosensitization was allowed) or thalidomide and its derivative treatments;
* Take VEGFR-TKI within 1 month, such as vandetanib, cabozantinib, lenvatinib, sunitinib and sorafenib;
* Allergic to apainib;
* Uncontrolled high blood pressure and heart disease;
* Patients with gastrointestinal bleeding risk;
* Coagulation disorders(INR>1.5×ULNAPTT>1.5×ULN);
* Uroprotein positive (Uroprotein≥2+ or 24-hour urinary protein quantity >1.0g);
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3-year
  The time from date of randomization until date of first documented disease progression or death from any cause

SECONDARY OUTCOMES:
Short-term treatment response rate | Three months after completion of the therapy
  Number of participants responded to the therapy according to RECIST 1.1
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Time to Response | From the initial treatment to first response, up to 3 years
  Time to first response to the therapy according to RECIST 1.1
Duration of Response | From first response to disease progression, up to 3 years
  Time from the first response to the therapy to disease progression
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v4.03 | Time interval from start to 3 months after completion of the therapy
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China